CLINICAL TRIAL: NCT06658691
Title: Multidisciplinary Approach in Tertiary Teaching Settings to Improve Diabetic Foot Care: an Investigation of Clinical and Economic Outcomes
Brief Title: Multidisciplinary Approach to Improve Diabetic Foot Care: an Investigation of Clinical and Economic Outcomes.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Jordan (Other)
Collaborators: Jordan University Hospital (Other)
Responsible Party: Principal Investigator, Majed Shafaamri, Clinical Research Assistant, University of Jordan
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 14296
Record Dates: First submitted 2024-10-19; First posted 2024-10-26 (Actual); Last update posted 2024-10-26 (Actual); Status verified 2024-10

CONDITIONS: Multidisciplinary Approach; Clinical Pharmacists; Diabetic Foot Ulcer (DFU); Multidisciplinary Care Team; Diabetes; Economic Outcomes
Keywords: Multidisciplinary approach; Clinical pharmacists; Jordan; Jordan University Hospital; Diabetic Foot Ulcer (DFU); Multidisciplinary team; Diabetes; Economic outcomes
MeSH Terms: conditions — Diabetic Foot; Diabetes Mellitus

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control group (No Intervention): Patients did not receive multidisciplinary approach
- Intervention group (Experimental): Patients received multidisciplinary approach
  Interventions: Other: Multidisciplinary approach

INTERVENTIONS:
Other: Multidisciplinary approach — The study investigated a multidisciplinary approach consisting of an endocrinologist, a diabetes specialized nurse, and a clinical pharmacist to assess and improve diabetic foot care by systematic screening, patients' risk categorization, therapy optimization, and tailored education.
  Risk of Diabetic Foot Ulcer (DFU) occurrence was assessed and evaluated by the endocrinologist, and the nurse based on the 2019 International Working Group on Diabetes Mellitus (IWGDF). At that point, only the clinical pharmacist knew about patients' allocations.
  According to risk stratification, the clinical pharmacist provided intervention patients with educational sessions and tailored materials during scheduled three months follow-up interviews at Jordan University Hospital (JUH) DFU-related clinics.
  Moreover, the study evaluated the impacts of the multidisciplinary approach on health-related Quality of Life (QoL) at baseline and at the end of the study. Economic impacts were also further analyzed.
  Arms: Intervention group

SUMMARY:
The study intervention was applying multidisciplinary approach consisting of an endocrinologist, a diabetes specialized nurse, and a clinical pharmacist to assess and improve diabetic foot care using a systematic screening, patients' risk categorization, therapy optimization, and tailored education.

DETAILED DESCRIPTION:
This is a single-blinded Randomized Controlled trial (RCT) study involving diabetic patients with (T1DM) and (T2DM) attending endocrine/diabetes, as well as, diabetic foot specialized surgery clinics for routine follow-ups at Jordan University Hospital (JUH) between 17 July 2022 and 30 Dec 2022.

The study evaluated the impacts of multidisciplinary approach in improving diabetic foot care. The clinical pharmacist role was to assess disease control, and to identify patients' therapeutic and educational needs through well-structured three months follow-up interviews with patients and/or their family members.

Moreover, the study investigated the impacts of multidisciplinary approach on health-related Quality of Life (QoL) at baseline and at the end of the study. Economic outcomes were also investigated relating to hospitalizations, length of stay, and cost of treatments.

The control group received standard care by hospital staff.

ELIGIBILITY:
Inclusion Criteria:

* Aged above 18 years old.
* Diabatic patients with T1DM and T2DM attending endocrine/diabetic and/or diabetic foot specialized surgery clinics for routine follow-ups at Jordan University Hospital (JUH).
* Diabetic patients with or without previous Diabetic Foot Ulcers (DFUs) and/or amputation.

Exclusion Criteria:

* Patients who were attending the clinics at the time of recruitment with active diabetic foot lesions and/or ulcers.
* Patients who were taking corticosteroid medications.
* Patients who were admitted to the hospital (inpatient admissions).
* Pregnant women attending gestational DM clinics.
* Patients with cognitive impairments and/or incapable to provide consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 119 (Actual)
Dates: Start 2022-07-17 (Actual); Primary Completion 2022-12-30 (Actual); Study Completion 2022-12-30 (Actual)

PRIMARY OUTCOMES:
Meeting the glycemic control goals | Up to 3 months
  In both study groups, the glycemic control outcomes were measured based on the percentage of patients meeting the HbA1c of less than 7%, and percentage of patients meeting Random Blood Sugar (RBS) of less than 180 mg/dl (ADA, 2018).

OTHER OUTCOMES:
Mean HbA1c | Up to 3 months
  In both study groups, the number of patients per each risk group was assessed. Across the study period, any disease progressions and/or improvements were also recorded, and mean HbA1c was measured.
Changes in Diabetic Foot Ulcer (DFU) predictors | Up to 3 months
  In both study groups, the number of patients per each risk group was assessed. Across the study period, any disease progressions and/or improvements were also recorded, and changes in Diabetic Foot Ulcer (DFU) predictors were measured.
Pharmacist interventions in identifying and resolving Treatment Related Problems (TRPs) | Up to 3 months
  Treatment related Problems (TRPs) were categorized into: unnecessary drug therapy, untreated conditions that require drug therapy, efficacy, safety, inappropriate knowledge, inappropriate adherence, and need for additional/more frequent drug monitoring.
  After identifying TRPs, the frequencies of TRPs were calculated within both study groups. The clinical pharmacist's recommendations were successfully delivered to the medical team, and all actions were documented.
  The rate at which the physician approved or rejected the recommendations was recorded, alongside the reason(s) was/were also examined.
Prevention of Diabetic Foot Ulcer (DFU) and/or amputation | Up to 3 months
  Intervention group was provided with targeted educational sessions in systematic, thorough, and repeated ways via face-to-face interviews, brochures, and recorded videos describing Diabetic Foot Ulcer (DFU) etiology, and daily foot self-care measures for patients and/or their family members. Also, the clinical pharmacist solved Treatment Related Problems (TRPs).
  Number of patients who developed newly DFUs events during the study period was assessed in both study groups.
Health-related Quality of Life (QoL) status | Up to 3 months
  The health-related Quality of Life (QoL) was assessed using EuroQol-5 Dimensions- 3 Levels (EQ-5D-3L) instrument, which included five aspects (Mobility, Self-care, Usual activities, Pain/ Discomfort, Anxiety/ Depression) at baseline, and at the end of the study for both study groups.
  The degree of severity of the EQ-5D-3L status was categorized based on Tongsiri and Cairns 2011 classification as mild, moderate, or severe.

CONTACTS AND LOCATIONS:
Overall Officials: Eman A Hammad, Principal Investigator — Department of Biopharmaceutics and Clinical Pharmacy, School of Pharmacy, University of Jordan
Locations (1):
- University of Jordan, Amman, Jordan